CLINICAL TRIAL: NCT02060149
Title: The Effect of Nebulization of Alkaline Solution on Treating Extensively Drug Resistant A. Baumannii Pneumonia With Cefoperazone and Sulbactam Plus Minocycline: A Multi-center Randomized Study
Brief Title: The Effect of Nebulization of Alkaline Solution on Treating XDRAB Pneumonia With C/S Plus Minocycline
Acronym: NAEDRAP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, songlq, vice director of department of respiratory and criticle care medicine, Xijing Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: xjhx-song1
Record Dates: First submitted 2013-03-10; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Pneumonia
Keywords: Extensively Drug Resistant A. Baumannii
MeSH Terms: conditions — Pneumonia | interventions — Minocycline; Cefoperazone; Sulbactam; Injections; Sodium Bicarbonate; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- no nebulization (Sham Comparator): Antibiotics protocol is C/S plus minocycline. That is Cefoperazone/ sulbactam 3.0g（intravenous infusion, q8h or q6h) combined with minocycline doxycycline 100mg (oral,q12h).No nebulization will given to these patients.
  Interventions: Drug: C/S plus minocycline.; Drug: No nebulization
- nebulization with pH 7.4 solution (Active Comparator): Patients will received the same antibiotics protocol with C/S plus minocycline and nebulization with pH 7.4 solution(Each time the volume of aerosol solution is 5ml, q8h).
  Interventions: Drug: C/S plus minocycline.; Drug: nebulization with pH 7.4 solution
- nebulization with pH 7.8 solution (Experimental): Patients will received the same antibiotics protocol with C/S plus minocycline and nebulization with pH 7.8 solution(Each time the volume of aerosol solution is 5ml, q8h).
  Interventions: Drug: C/S plus minocycline.; Drug: nebulization with pH 7.8 solution

INTERVENTIONS:
Drug: C/S plus minocycline. — Cefoperazone/ sulbactam 3.0g（intravenous infusion, q8h or q6h) combined with minocycline doxycycline 100mg (oral, q12h).
  Other Names: CEFOPERAZONE SODIUM AND SULBACTAM SODIUM FOR INJECTION
Drug: nebulization with pH 7.4 solution — Patients will receive the nebulization with Sodium Bicarbonate of pH 7.4 (Each time the volume of aerosol solution is 5ml, q8h).
  Other Names: Sodium Bicarbonate
  Arms: nebulization with pH 7.4 solution
Drug: nebulization with pH 7.8 solution — Patients will receive the nebulization with Sodium Bicarbonate of pH 7.8 (Each time the volume of aerosol solution is 5ml, q8h).
  Other Names: Sodium Bicarbonate
  Arms: nebulization with pH 7.8 solution
Drug: No nebulization — No nebulization will be given to the patients.
  Other Names: sham
  Arms: no nebulization

SUMMARY:
The mortality of pneumonia with extensively drug resistant Acinetobacter baumannii (XDRAB) is still high, even if these patients received certain strong anti-infection treatment such us the combination of cefoperazone-sulbactam (C/S) and minocycline. Health airway lining fluid is mildly alkaline but airway acidification usually appears for the infection of XDRAB. The hypothesis is offered that the biologic activity of XDRAB might be inhibited if the circumstance including pH is changed. In the vitro study we observed that the inhibit effect of antibiotics on XDRAB growth was improved significantly by alkaline solution within the scope of physiology. So the aim of this clinical study is to explore the effects of nebulization of alkaline Solution on C/S plus minocycline on the pneumonia with XDRAB.

DETAILED DESCRIPTION:
Pneumonia patients with XDRAB are eligible for this multicenter study, do not meet the exclusion criteria and will sign the informed consent. They will received the anti-infection protocol with Cefoperazone/ sulbactam 3.0g（intravenous infusion, q8h or q6h) combined with minocycline doxycycline 100mg (oral, q12h). All enrolled patients were randomly divided into three groups according to the difference in pH value of aerosol inhalation with sodium bicarbonate solution. Group one is blank-control and patients will received usual antibiotic treatment without inhalation. The pH value in group two is 7.4 and that in group is 7.8. Each time the volume of aerosol solution is 5ml, q8h. The average course of treatment will be two weeks. Clinical indexes will be collected including vital signs, pulmonary rales, cough level, expectoration level, sputum color,blood count, arterial blood gas, biochemical parameters, chest X-ray score, APACHE II score, clinical pulmonary infection score, ECG, sputum culture, et al.The primary endpoints are pathogenic clearance rate and recovery rate. The secondary end point is adverse reaction rate.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years old, male or female
* The pneumonia patients met the diagnostic criteria, and clinical pulmonary infection score (CPIS) ≥ 5;
* The sputum bacteriology detection only prompted Acinetobacter baumannii culture for pathogens concentration meets the diagnostic criteria of the Chinese hospital-acquired pneumonia diagnosis and treatment guidelines, 2002 edition of "Acinetobacter baumannii and susceptibility results show only 1 to 2 sensitive to antimicrobial drugs (polymyxin, minocycline or tegafur doxycycline);
* Cephalosporins or tetracyclines drug treatment without a history of allergies and contraindications;
* Be able to accept inhalation therapy.
* Informed consent gained

Exclusion Criteria:

* Refused to accept inhalation therapy
* Renal insufficiency, creatinine clearance (Cockcroft-Gault formula) (CLcr) 15 ml / min or less;
* Liver dysfunction, defined as Child-Pugh score B or C
* Within one week before the start of cefoperazone sulbactam, minocycline treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Pathogenic Clearance rate and recovery rate | one treatment course for about two weeks

SECONDARY OUTCOMES:
adverse reaction rate | one treatment course for about two weeks

OTHER OUTCOMES:
hospital time and mortality | about four weeks

CONTACTS AND LOCATIONS:
Overall Officials: liqiang song, doctor, Principal Investigator — first affiliated hospital, fourth military medical university
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China